CLINICAL TRIAL: NCT04264208
Title: Evaluation of Patients With Low-Risk and Intermediate-Risk Prostate Cancer Scheduled for High-Dose Rate Brachytherapy Using 68-Ga-RM2 PET, 68Ga-PSMA-11 PET and Multi Parametric MRI
Brief Title: HDR Brachytherapy 68-Ga-RM2 PET, 68-Ga-PSMA-11 PET &Multi Parametric MRI in Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual due to pandemic and logistics
Sponsor: Andrei Iagaru (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Andrei Iagaru, Professor of Radiology (Nuclear Medicine), Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB-51987; PROS0098 (Other: OnCore); NCI-2020-02779 (Registry Identifier: CTRP); 1R01CA230438 (NIH)
Record Dates: First submitted 2020-02-04; First posted 2020-02-11 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — BAY 86-7548; gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 68Ga-RM2 PET MRI then 68 Ga PMSA11 PET/MRI (Experimental): Subjects will undergo either 68Ga RM2 PET/MRI followed within 2 weeks by 68Ga PMSA11 PET/MRI. Two x intravenous (IV) 68Ga-RM2 PET/MRI with a 68Ga dosage of 140 mBq (3.8 mCi), +/- 20%, Two x intravenous (IV) 68Ga-PMSA11 PET/MRI with a 68Ga dosage of 111 to 259 mBq (3 to 7 mCi)
  Interventions: Drug: 68-Ga RM2.; Drug: 68-Ga PSMA11; Device: PET/MRI
- 68Ga-PSMA-11 PET MRI then 68Ga-RM2 PET MRI (Experimental): Subjects will undergo 68Ga PMSA11 PET/MRI followed within 2 weeks by 68Ga RM2 PET/MRI. Two x intravenous (IV) 68Ga-RM2 PET/MRI with a 68Ga dosage of 140 mBq (3.8 mCi), +/- 20%, Two x intravenous (IV) 68Ga-PMSA11 PET/MRI with a 68Ga dosage of 111 to 259 mBq (3 to 7 mCi)
  Interventions: Drug: 68-Ga RM2.; Drug: 68-Ga PSMA11; Device: PET/MRI

INTERVENTIONS:
Drug: 68-Ga RM2. — PET radiopharmaceutical
  Other Names: BAY86 7548; 68Ga DOTA Bombesin
Drug: 68-Ga PSMA11 — PET radiopharmaceutical
  Other Names: DFKZ 11; HBED CC PSMA; Heidelberg compound
Device: PET/MRI — PET/MR scanner by GE healthcare
  Other Names: PET/MR scanner

SUMMARY:
This study is being conducted to determine whether the combination of imaging agents 68-Ga RM2 and 68-Ga PMSA11 is better at assessing response to high dose rate (HDR) local therapy than standard imaging or biopsy in patients with known prostate cancer (PC)

DETAILED DESCRIPTION:
Primary Objective:

1. To demonstrate that 68Ga-RM2 and 68Ga-PSMA-11 PET/MRI can detect additional cancers over mpMRI.
2. To demonstrate that 68Ga-RM2 and 68Ga-PSMA-11 PET/MRI can assess changes in response to treatment and predict progression free survival (PFS) at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age;
* Patients must be able to provide informed consent;
* Histologically proven low-grade or intermediate-grade prostate cancer (PC)
* Scheduled to undergo targeted local therapy (HDR brachytherapy).

Exclusion Criteria:

* Inability to lie still for the entire imaging time;
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.);
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance;
* Metallic implants (contraindicated for MRI).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 4 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei H Iagaru, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Cancer Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants signed consent and three participants were randomized to treatment.
Groups:
- 68Ga-RM2 PET MRI Then 68Ga PSMA 11 PET/MRI: Subjects will undergo either 68Ga RM2 PET/MRI followed within 2 weeks by 68Ga PSMA 11 PET/MRI.
- 68Ga-PSMA-11 PET MRI Then 68Ga-RM2 PET MRI: Subjects will undergo 68Ga PSMA 11 PET/MRI followed within 2 weeks by 68Ga RM2 PET/MRI.
Period: Pre-HDR Scan Sequence
Arm/Group | 68Ga-RM2 PET MRI Then 68Ga PSMA 11 PET/MRI | 68Ga-PSMA-11 PET MRI Then 68Ga-RM2 PET MRI
Started | 1 | 2
Received First Scan in Sequence | 1 | 2
Received Second Scan in Sequence | 0 | 1
Completed | 1 | 2
Not Completed | 0 | 0
Period: HDR Treatment at 2 Months
Arm/Group | 68Ga-RM2 PET MRI Then 68Ga PSMA 11 PET/MRI | 68Ga-PSMA-11 PET MRI Then 68Ga-RM2 PET MRI
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0
Period: Post-HDR Scan Sequence at 10 Months
Arm/Group | 68Ga-RM2 PET MRI Then 68Ga PSMA 11 PET/MRI | 68Ga-PSMA-11 PET MRI Then 68Ga-RM2 PET MRI
Started | 1 | 2
Received First Scan in Sequence | 0 | 1
Received Second Scan in Sequence | 0 | 1
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 68Ga-RM2 PET MRI Then 68Ga PSMA 11 PET/MRI: Subjects will undergo either 68Ga RM2 PET/MRI followed within 2 weeks by 68Ga PSMA11 PET/MRI.
- Total: Total of all reporting groups
Arm/Group | 68Ga-RM2 PET MRI Then 68Ga PSMA 11 PET/MRI | 68Ga-PSMA-11 PET MRI Then 68Ga-RM2 PET MRI | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Assessment of PET Based PC Lesions
Description: Assessment of whether 68-Ga-RM2 and 68-Ga-PSMA-11 PET/MRI can detect additional cancers over mpMRI. Detection of PC lesions will be assessed by 68Ga PSMA11 and 68Ga RM2 PET scans.
Time Frame: Day 1 (first scan) and 2 weeks (second scan) relative to baseline. First scan was approximately 2 months prior to HDR treatment
Population: Participants with pre HDR treatment scan data
Measure: Count of Participants; unit: Participants
Groups:
- 68Ga-RM2 PET MRI: Subjects receive 68Ga RM2 PET/MRI.
- 68Ga-PSMA-11 PET MRI: Subjects receive 68Ga PSMA11 PET/MRI.
Arm/Group | 68Ga-RM2 PET MRI | 68Ga-PSMA-11 PET MRI
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

2. Primary Outcome: Number of Participants for Which an Assessment of PET Based Therapeutic Response to HDR is Successfully Obtained
Description: Assessment of whether 68Ga-RM2 and 68Ga-PSMA-11 PET/MRI can assess changes in response to treatment. Therapeutic response to HDR will be assessed by 68Ga PSMA 11 and 68Ga RM2 PET scans. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: as for outcome 1
Population: Participants who received post HDR scan
Measure: Count of Participants; unit: Participants
Arm/Group | 68Ga-RM2 PET MRI | 68Ga-PSMA-11 PET MRI
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

3. Primary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) will be assessed as survival without progression at 24 months. The outcome is reported as the number (without dispersion) of the participants alive without progression.
Time Frame: 24 months
Population: No participant had month 24 data (all discontinued prior)
Arm/Group | 68Ga-RM2 PET MRI | 68Ga-PSMA-11 PET MRI
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 13 months
Arm/Group | 68Ga-RM2 PET MRI | 68Ga-PSMA-11 PET MRI
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
Early termination led to a small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT04264208/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT04264208/ICF_002.pdf